CLINICAL TRIAL: NCT01846520
Title: A Randomized Trial of a Family Caregiver Palliative Care Intervention
Brief Title: Family Caregiver Palliative Care Intervention in Supporting Caregivers of Patients With Stage II-IV Gastrointestinal, Gynecologic, Urologic and Lung Cancers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); American Cancer Society (ACS) National Office (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 08176; NCI-2013-00839 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-05-01; First posted 2013-05-03 (Estimated); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Healthy Subject; Localized Transitional Cell Cancer of the Renal Pelvis and Ureter; Metastatic Transitional Cell Cancer of the Renal Pelvis and Ureter; Psychosocial Effects of Cancer and Its Treatment; Recurrent Bladder Cancer; Recurrent Cervical Cancer; Recurrent Colon Cancer; Recurrent Gastric Cancer; Recurrent Ovarian Epithelial Cancer; Recurrent Ovarian Germ Cell Tumor; Recurrent Pancreatic Cancer; Recurrent Rectal Cancer; Recurrent Renal Cell Cancer; Recurrent Transitional Cell Cancer of the Renal Pelvis and Ureter; Recurrent Urethral Cancer; Recurrent Uterine Sarcoma; Regional Transitional Cell Cancer of the Renal Pelvis and Ureter; Stage II Bladder Cancer; Stage II Renal Cell Cancer; Stage II Urethral Cancer; Stage IIA Cervical Cancer; Stage IIA Colon Cancer; Stage IIA Gastric Cancer; Stage IIA Ovarian Epithelial Cancer; Stage IIA Ovarian Germ Cell Tumor; Stage IIA Pancreatic Cancer; Stage IIA Rectal Cancer; Stage IIA Uterine Sarcoma; Stage IIB Cervical Cancer; Stage IIB Colon Cancer; Stage IIB Gastric Cancer; Stage IIB Ovarian Epithelial Cancer; Stage IIB Ovarian Germ Cell Tumor; Stage IIB Pancreatic Cancer; Stage IIB Rectal Cancer; Stage IIB Uterine Sarcoma; Stage IIC Colon Cancer; Stage IIC Ovarian Epithelial Cancer; Stage IIC Ovarian Germ Cell Tumor; Stage IIC Rectal Cancer; Stage III Bladder Cancer; Stage III Pancreatic Cancer; Stage III Renal Cell Cancer; Stage III Urethral Cancer; Stage IIIA Cervical Cancer; Stage IIIA Colon Cancer; Stage IIIA Gastric Cancer; Stage IIIA Ovarian Epithelial Cancer; Stage IIIA Ovarian Germ Cell Tumor; Stage IIIA Rectal Cancer; Stage IIIA Uterine Sarcoma; Stage IIIB Cervical Cancer; Stage IIIB Colon Cancer; Stage IIIB Gastric Cancer; Stage IIIB Ovarian Epithelial Cancer; Stage IIIB Ovarian Germ Cell Tumor; Stage IIIB Rectal Cancer; Stage IIIB Uterine Sarcoma; Stage IIIC Colon Cancer; Stage IIIC Gastric Cancer; Stage IIIC Ovarian Epithelial Cancer; Stage IIIC Ovarian Germ Cell Tumor; Stage IIIC Rectal Cancer; Stage IIIC Uterine Sarcoma; Stage IV Bladder Cancer; Stage IV Gastric Cancer; Stage IV Ovarian Epithelial Cancer; Stage IV Ovarian Germ Cell Tumor; Stage IV Pancreatic Cancer; Stage IV Renal Cell Cancer; Stage IV Urethral Cancer; Stage IVA Cervical Cancer; Stage IVA Colon Cancer; Stage IVA Rectal Cancer; Stage IVA Uterine Sarcoma; Stage IVB Cervical Cancer; Stage IVB Colon Cancer; Stage IVB Rectal Cancer; Stage IVB Uterine Sarcoma; Ureter Cancer; Stage IIA Lung Carcinoma; Stage IIB Lung Carcinoma; Stage IIIA Lung Carcinoma; Stage IIIB Lung Carcinoma
MeSH Terms: conditions — Urinary Bladder Neoplasms; Uterine Cervical Neoplasms; Colonic Neoplasms; Stomach Neoplasms; Carcinoma, Ovarian Epithelial; Pancreatic Neoplasms; Rectal Neoplasms; Carcinoma, Renal Cell; Urethral Neoplasms; Ureteral Neoplasms; Lung Neoplasms | interventions — Early Intervention, Educational; Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (FCPCI) (Experimental): Participants receive FCPCI with an APN, comprising 4 home education sessions once weekly followed by 4 telephone support sessions for 30 minutes once monthly and 24 hour telephone support available for 6 months.
  Interventions: Other: educational intervention; Behavioral: telephone-based intervention; Procedure: quality-of-life assessment; Other: questionnaire administration
- Arm II (usual care) (No Intervention): Participants receive usual care.

INTERVENTIONS:
Other: educational intervention — Receive FCPCI home education sessions
  Other Names: intervention, educational
  Arms: Arm I (FCPCI)
Behavioral: telephone-based intervention — Receive FCPCI telephone support sessions and 24 hour telephone support
  Arms: Arm I (FCPCI)
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
  Arms: Arm I (FCPCI)
Other: questionnaire administration — Ancillary studies
  Arms: Arm I (FCPCI)

SUMMARY:
This randomized clinical trial studies the Family Caregiver Palliative Care Intervention in supporting caregivers of patients with stage II-IV gastrointestinal, gynecologic, urologic and lung cancers. Education and telephone counseling may reduce stress and improve the well-being and quality of life of caregivers of cancer patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. Test the effects of the Family Caregiver Palliative Care Intervention (FCPCI) on family caregivers of patients with gastrointestinal, gynecologic, urologic and lung cancers in the experimental group on caregiver burden and caregiving skills preparedness as compared to family caregivers in the control group.

II. Test the effects of the FCPCI on family caregivers of patients with gastrointestinal, gynecologic, urologic and lung cancers in the experimental group on quality of life (QOL) and psychological distress as compared to family caregivers in the control group.

SECONDARY OBJECTIVES: I. Describe family caregivers' self-care behavior, comparing the experimental and control groups.

II. Describe family caregivers' resource use, comparing the experimental and control groups.

III. Identify subgroups of family caregivers who benefit most from the FCPCI in relation to sociodemographic, health status, and patient characteristics.

IV. Describe family caregivers' satisfaction with the FCPCI.

V. Describe caregiver out-of-pocket costs and the cost of the intervention.

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I: Participants receive FCPCI with an advanced practice nurse (APN), comprising 4 home education sessions once weekly followed by 4 telephone support sessions for 30 minutes once monthly and 24 hour telephone support available for 6 months.

ARM II: Participants receive usual care

ELIGIBILITY:
Inclusion Criteria:

* Primary family caregivers of cancer patients with gastrointestinal (colorectal, pancreatic, gastric), gynecologic, urinary or lung cancers who are entering the City of Hope for treatment or follow-up
* Primary family caregivers of cancer patients who are diagnosed with stage II-IV disease
* Primary family caregivers of cancer patients with > 6 months prognosis
* Living within a 50 mile radius of the City of Hope

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-10; Primary Completion 2019-05-23 (Actual); Study Completion 2019-05-23 (Actual)

PRIMARY OUTCOMES:
Effects of Family Caregiver Palliative Care Intervention (FCPCI) on caregiver burden | Up to 6 months
  Analysis of covariance (ANCOVA) will be used to test group differences. Caregiver burden subscales may be tested using multivariate ANCOVA (MANCOVA).
Effects of FCPCI on caregiving skills preparedness | Up to 6 months
  ANCOVA will be used to test group differences. Caregiver burden subscales may be tested using MANCOVA.
Effects of FCPCI on Quality Of Life (QOL) | Up to 6 months
  ANCOVA will be used to test group differences. MANCOVA may be used to test group differences of QOL subscale scores.
Effects of FCPCI on psychological distress | Up to 6 months
  ANCOVA will be used to test group differences. MANCOVA may be used to test group differences of QOL subscale scores.

SECONDARY OUTCOMES:
Caregiver's self-care behavior | Up to 6 months
  Qualitative analyses will be conducted on the narrative responses to the Self-Care Behaviors instrument. Self-care behaviors will be coded within each category. Results will be reviewed for consensus and validation, and any discrepancies will be resolved. Tables of coded themes with examples will be created.
Caregivers' resource use | Up to 6 months
  The qualitative analysis will be conducted on the narrative responses to the Resource Use instrument. Resources will be coded within each category. Results will be reviewed for consensus and validation, and any discrepancies will be resolved. Tables of categories and codes will be created.
Identification of subgroups of family caregivers who benefit most from the FCPCI in relation to sociodemographic, health status, and patient characteristics | 3 months
  In four separate hierarchical multiple linear regression analyses, the 3 month outcome measure (caregiver burden, skills preparedness, psychological distress, and total QOL) will be regressed first on baseline measures for the relevant outcomes, followed by demographic and caregiver health status variables, and then by patient characteristics and severity of illness, using dummy-coding as appropriate.
Family caregivers' satisfaction with the FCPCI | 6 months
  A descriptive analysis of the brief satisfaction survey item results for subjects in the experimental group will be conducted, summarizing number and percent for normal data or means and standard deviations for continuous data.
Caregiver out-of-pocket costs | Up to 6 months
  A descriptive analysis of family caregivers' costs will be conducted.

CONTACTS AND LOCATIONS:
Overall Officials: Betty Ferrell, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States